CLINICAL TRIAL: NCT05558579
Title: Comparison of Postoperative Sling Use in Patient Outcomes After Isolated Biceps Tenodesis
Brief Title: Use of Postop Sling After Biceps Tenodesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Michael Karns, MD., Assistant Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20220856
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Biceps Tenodesis
Keywords: shoulder rehabilitation; shoulder sling; biceps disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Using Sling (No Intervention): Patients will continue using shoulder sling per standard of care
- Patients Without Sling (Experimental): Patients will not use shoulder sling postoperatively.
  Interventions: Other: No sling use

INTERVENTIONS:
Other: No sling use — Patients will not use standard of care sling
  Arms: Patients Without Sling

SUMMARY:
The purpose of this study is to evaluate whether the use of a sling after surgery (biceps tenodesis) is required in recovery and rehabilitation. Biceps tenodesis is one of the most common surgeries for patients who have biceps tendon inflammation and/or instability, rotator cuff tears, and labral tears that do not get better with medications or physical therapy. A biceps tenodesis involves cutting the biceps tendon and reconnecting it to the shoulder with sutures or metal screws. After surgery, most patients are required to wear a shoulder sling and limit certain arm motions to protect the healing tendon. A recent study found using a more flexible rehabilitation protocol for biceps tenodesis did not change outcomes (strength or range-of-motion) and allows patients to return to some regular activities earlier. This data suggests patients may not need to wear a sling after surgery. Therefore, this study aims to evaluate this.

This study will have two groups-one that continues to wear the sling, and one that does not. Patients will be randomly assigned to one of these groups. At each follow-up visit after surgery, shoulder strength and range-of-motion will be measured and several surveys about shoulder function will be completed. These surveys will provide information to compare between both groups. If assigned to the group that wears the sling, patients will record how often they are wearing the sling in a paper diary/log. Additionally, at the 6-month follow-up, an ultrasound will be obtained to make sure the tendon is healing properly regardless of which group patients are assigned to. Finally, medical history will be collected to identify protective and risk factors for any differences that might be found.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo open or arthroscopic isolated BT for diagnoses including but not limited to biceps tendinitis or tenosynovitis, biceps tendon tears, partial-thickness rotator cuff tears, subacromial bursitis, superior labrum from anterior to posterior (SLAP) tear, biceps instability
* Patients with minimum 6-month follow-up

Exclusion Criteria:

* Patients who undergo any concomitant procedures necessitating ROM restrictions, including but not limited to rotator cuff repair, labral repair, SLAP lesion repair, or shoulder arthroplasty
* Patients with history of prior ipsilateral proximal biceps procedures
* Patients with history of conditions resulting in severe shoulder strength and ROM limitations (e.g. severe degenerative glenohumeral osteoarthritis, polymyalgia rheumatica, cervical radiculopathy, significant muscle paralysis, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
Percent of Complications As Measured by Medical Records | Up to 2 years
Degrees of Range-of-Motion As Measured by Physical Exam | Up to 30 minutes
Strength as Measured by Physical Exam | Up to 30 minutes
  Strength is measured on a 5-point scale with 0 being no discernible muscle contraction and 5 being muscle contraction and maximum resistance

SECONDARY OUTCOMES:
Pain as Measured by the Visual Analog Scale | Up to 5 minutes
  VAS is a 10-point scale with 0 being no pain and 10 being worst possible pain
Shoulder Function as Measured by the American Shoulder and Elbow Surgeons (ASES) | Up to 15 minutes
  ASES is a 17-item survey that has a score from 0-100
Shoulder Function as Measured by the Simple Shoulder Test (SST) | Up to 15 minutes
  SST is a 12-item survey that has a score up to 12 points
Shoulder Function as Measured by Constant Murley Score (CMS) | Up to 15 minutes
  CMS is scored up to 100 points maximum
Shoulder Function as Measured by the Western Ontario Rotator Cuff (WORC) Index | Up to 15 minutes
  WORC is a 21-item survey scored on a scale from 2,100 to 0
Shoulder Function as Measured by the Single Assessment Numeric Evaluation (SANE) | Up to 5 minutes
  SANE is a 1-item survey that has a score from 0-100
Percent of Patients Satisfied as Measured by Patient Survey | Up to 5 minutes
  Yes/no survey asking about satisfaction with care

CONTACTS AND LOCATIONS:
Overall Officials: Michael Karns, MD, Principal Investigator — University Hospitals; Kallie Chen, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No